CLINICAL TRIAL: NCT04827472
Title: A Randomized, Double Blind, Placebo-controlled, Single Dose, Dose-escalation Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Pharmacodynamics After Intravenous DWJ1521 Administration in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Pharmacodynamics After Intravenous DWJ1521 Administration in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1521101
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution; fexuprazan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part1(Cohort1) : DWJ1521 Amg (Experimental)
  Interventions: Drug: Normal saline; Drug: DWJ1521
- Part1(Cohort2) : DWJ1521 Bmg (Experimental)
  Interventions: Drug: Normal saline; Drug: DWJ1521
- Part1(Cohort3) : DWJ1521 Cmg (Experimental)
  Interventions: Drug: Normal saline; Drug: DWJ1521
- Part1(Cohort4) : DWJ1521 Dmg (Experimental)
  Interventions: Drug: Normal saline; Drug: DWJ1521
- Part2 : DWJ1521 Xmg (Experimental)
  Interventions: Drug: DWJ1521
- Part2 : DWP14012 Tablet (Experimental)
  Interventions: Drug: DWP14012 Tablet

INTERVENTIONS:
Drug: Normal saline — 100ml
  Arms: Part1(Cohort1) : DWJ1521 Amg; Part1(Cohort2) : DWJ1521 Bmg; Part1(Cohort3) : DWJ1521 Cmg; Part1(Cohort4) : DWJ1521 Dmg
Drug: DWJ1521 — Single dose
  Arms: Part1(Cohort1) : DWJ1521 Amg; Part1(Cohort2) : DWJ1521 Bmg; Part1(Cohort3) : DWJ1521 Cmg; Part1(Cohort4) : DWJ1521 Dmg; Part2 : DWJ1521 Xmg
Drug: DWP14012 Tablet — Single dose, Tablet
  Arms: Part2 : DWP14012 Tablet

SUMMARY:
The safety/tolerability and pharmacokinetic properties of DWJ1521 are evaluated after single intravenous administration of DWJ1521 in healthy adults.

The safety/tolerability and pharmacokinetic properties of DWJ1521 single intravenous administration and DWP14012 single oral administration in healthy adults are compared.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 50 years old at the time of screening test
2. Those who weigh 55.0 kg or more and 90.0 kg or less at the time of the screening test and have a body mass index (BMI) of 18.0 or more and 28.0 or less ☞ BMI(kg/m2) = weight(kg) / {height(m)}2

Exclusion Criteria:

1. Clinically significant, liver, kidney, nervous system, immune system, respiratory system, endocrine system, etc., or blood or tumor disease, cardiovascular disease, mental disease (mood disorder, obsessive-compulsive disorder, etc.) or have a history of character
2. Those with a history of gastrointestinal diseases (gastrointestinal ulcers, gastritis, gastric cramps, gastroesophageal reflux disease, Crohn's disease, etc.) that may affect the safety and pharmacokinetics evaluation of investigational drugs, and those with a history of gastrointestinal surgery (However, simple appendic surgery and hernia surgery are excluded)
3. Those who were tested positive for Helicobacter pylori
4. serologic test results (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test) positive
5. Those whose blood AST and ALT exceeds 1.5 times the upper limit of the normal range in screening tests including additional tests.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
24h pH monitoring, the ratio of the time remaining above pH 4, 6 (time%) | [Time Frame: [Time Frame: 0 - 72 hours after dosing]]

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea